CLINICAL TRIAL: NCT00931801
Title: A Pilot Study of the Novel Antiretroviral Combination of Atazanavir and Raltegravir in HIV-1 Infected Subjects With Virologic Suppression on a Standard Regimen of Boosted Atazanavir, Tenofovir and Emtricitabine
Brief Title: BATAR: Individuals Currently Taking Boosted Atazanavir as Part of an HIV Treatment Regimen Will be Evaluated to See if Substituting Raltegravir for Nucleoside Transcriptase Inhibitors Will be Safe and Well Tolerated.
Acronym: BATAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Community Research Initiative of New England (Other)
Collaborators: Bristol-Myers Squibb (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-102
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: HIV
Keywords: AIDS; HIV; Atazanavir; Raltegravir; Tenofovir; protease inhibitors
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Atazanavir Sulfate; Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention Arm No.1 (Experimental)
  Interventions: Drug: atazanavir/raltegravir
- Intervention Arm No.2 (Experimental)
  Interventions: Drug: atazanavir/raltegravir
- Control Arm (Active Comparator): Continue baseline regimen
  Interventions: Drug: atazanavir/tenofovir/emtricitabine

INTERVENTIONS:
Drug: atazanavir/raltegravir — Atazanavir/r 300/100mg once daily plus raltegravir 400mg twice daily
  Arms: Intervention Arm No.1
Drug: atazanavir/raltegravir — Atazanavir 300mg twice daily plus raltegravir 400mg twice daily
  Arms: Intervention Arm No.2
Drug: atazanavir/tenofovir/emtricitabine — Continue baseline regimen of atazanavir/r 300/100mg once daily plus tenofovir and emtricitabine
  Other Names: Truvada
  Arms: Control Arm

SUMMARY:
The purpose of this Phase IV pilot study is to evaluate the safety, tolerability, and satisfaction of a nucleoside analog reverse-transcriptase inhibitors (NRTI)sparing regimen for participants fully suppressed on an atazanavir/ritonavir based highly active antiretroviral therapy (HAART)regimen plus emtricitabine/tenofovir (Truvada). Several pharmacologic factors support this concept including the favorable drug interaction between atazanavir and raltegravir. Participants will be randomized to either continue on their current regimen or one of two study arms (atazanavir 300mg plus ritonavir 100mg daily plus raltegravir 400mg twice daily or atazanavir 300mg twice daily plus raltegravir 400mg twice daily). Participants will be followed for 48 weeks for safety, tolerability, and satisfaction. After baseline, the participants will have six clinic visits for evaluation and labs.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Treatment with a stable antiretroviral regiment containing boosted atazanavir, tenofovir and emtricitabine at screen and for at least 90 days prior to screening
* No plan to make changes to HIV treatment regimen (other than those required by the study) in the next 48 weeks
* Undetectable HIV RNA at screening AND no HIV RNA>200 copies during the 180 day period prior to screening
* CD4 count>200
* No evidence of resistance to any of the drugs in any of the 3 arms, if prior resistance tests are available
* Subjects who, in the opinion of their treating physicians, would be candidates to switch antiretroviral medications
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of study drug
* Ability and willingness to provide written informed consent and comply with protocol requirements

Exclusion Criteria:

* Prior exposure to raltegravir or elvitegravir
* Women who are pregnant, breast-feeding, or with a positive pregnancy test
* Sexually active fertile men not using effective birth control if their female partners are of child-bearing potential
* Women of child-bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of study drug
* Life expectancy less than 6 months
* Presence of any currently active AIDS defining conditions with the exception of stable cutaneous Kaposi's sarcoma
* Treatment with proton-pump inhibitor or H2-receptor antagonist
* ECG demonstrating atrioventricular block, prolonged QRS interval greater than 12 ms, or known complete bundle branch block
* Acute or chronic hepatitis B infection as evidenced by presence of hepatitis B surface antigen and absence of hepatitis B surface antibody
* Clinical or laboratory evidence of significantly decreased hepatic function of decompensation irrespective of liver enzyme levels
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Calvin J Cohen, MD, MSc, Principal Investigator — Community Research Initiative
Locations (9):
- United States (9):
  - Spectrum Medical Group, Phoenix, Arizona
  - AIDS Healthcare Foundation, Los Angeles, California
  - Denver Public Health, Denver, Colorado
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - Orlando Immunology Center, Orlando, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Christi Research, Wichita, Kansas
  - Community Research Initiative of New England - Boston, Boston, Massachusetts
  - David M. Lee, MD, PA d/b/a/ Uptown Physicians' Group, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was initiated on 15 APR 2010 and enrolled subjects through 31 JAN 2011. Recruitment and screening took place at 10 participating sites (9 medical clinics and 1 clinical research organization). 43 subjects were enrolled.
Pre-assignment Details: There were 7 participants that did not meet eligibility criteria (either due to disallowed concomitant medication use or safety labs outside of the required parameters). 2 of those 7 subjects re-screened at a later date and were confirmed eligible. 2 subjects withdrew consent after the screening visit but prior to starting the assigned treatment.
Groups:
- Control Arm: atazanavir/tenofovir/emtricitabine : Continue baseline regimen of atazanavir/r 300/100mg once daily plus tenofovir and emtricitabine
- Intervention Arm No.1: atazanavir/raltegravir: switch to atazanavir/r 300/100mg once daily plus raltegravir 400mg twice daily
- Intervention Arm No.2: atazanavir/raltegravir: switch to atazanavir 300mg twice daily plus raltegravir 400mg twice daily
Period: Overall Study
Arm/Group | Control Arm | Intervention Arm No.1 | Intervention Arm No.2
Started | 14 | 15 | 14
Completed | 13 | 14 | 10
Not Completed | 1 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Confirmed Virologic Failure | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intervention Arm No.1 | Intervention Arm No.2 | Total
Number analyzed (Participants) | 14 | 15 | 14 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (11.6) | 47.6 (11.5) | 46.6 (6.6) | 45.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 12 | 13 | 13 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 5 | 13
  Not Hispanic or Latino | 8 | 13 | 9 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 9
  White | 9 | 12 | 11 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 14 | 43
Mean CD4 [Mean (Standard Deviation); unit: cells/mm3] | 544.6 (197.7) | 518.5 (198.9) | 533.9 (198.3) | 532.0 (193.8)

OUTCOME MEASURES:

1. Primary Outcome: Maintenance of Virologic Suppression
Description: To evaluate and compare maintenance of virologic suppression with raltegravir (RAL) 400mg 2x daily plus atazanavir (ATV) dosed either as ATV/ritonavir (RTV)300/100mg 1x daily or ATV 300mg 2x daily in subjects with virologic suppression on a standard regimen of ATV/RTV plus Truvada. Virologic suppression is defined as HIV RNA < 40 copies/mL.
Time Frame: 48 weeks
Population: All enrolled participants were included in this analysis of primary outcome measurement.
Measure: Number; unit: participants
Groups:
- Control Arm: Continue baseline regimen of atazanavir/ritonavir 300/100mg once daily plus tenofovir and emtricitabine
- Intervention Arm No.1: switch to atazanavir/ritonavir 300/100mg once daily plus raltegravir 400mg twice daily
- Intervention Arm No.2: switch to atazanavir 300mg twice daily plus raltegravir 400mg twice daily
Arm/Group | Control Arm | Intervention Arm No.1 | Intervention Arm No.2
Number analyzed (Participants) | 14 | 15 | 14
participants
  Virologic Response | 13 | 14 | 10
  Confirmed Virologic Failures | 0 | 0 | 3
  Withdrawal Due to AE; HIV RNA < 50 copies/mL | 0 | 0 | 1
  Other Withdrawal; HIV RNA < 50 copies/mL | 1 | 1 | 0

2. Secondary Outcome: The Difference in CD4 From Baseline to Week 48
Description: Change in mean CD4 from Baseline to Week 48.
Time Frame: Baseline and Week 48
Population: Values included for all enrolled participants excluding participants with confirmed virologic failure or those missing values due to early withdrawal, loss to follow-up or lab error.
Measure: Mean (Standard Deviation); unit: cells/mm3
Groups:
- Control Arm: Continue baseline regimen of atazanavir/r 300/100mg once daily plus tenofovir and emtricitabine
- Intervention Arm No.1: switch to atazanavir/r 300/100mg once daily plus raltegravir 400mg twice daily
- Total: All study arms combined
Arm/Group | Control Arm | Intervention Arm No.1 | Intervention Arm No.2 | Total
Number analyzed (Participants) | 12 | 14 | 10 | 36
cells/mm3
  CD4 at Baseline | 535.8 (210.9) | 514.1 (205.7) | 539.1 (206.2) | 528.3 (201.9)
  CD4 at Week 48 | 611.2 (218.1) | 526.3 (210.5) | 507.2 (201.7) | 549.3 (209.5)
  CD4 Change | 75.4 (133.9) | 12.1 (96.4) | -31.9 (122.0) | 21.0 (121.5)

3. Secondary Outcome: The Change in Adherence to Study Treatment Arm From Baseline to Week 48
Description: Adherence to study treatment reported as the percentage of doses of the prescribed treatment arm regimen taken, described by each subject through recall of dosing in the three days prior to the visit Baseline and Week 48 vistis. The change in adherence is reflected as the difference of the mean percentage of adherence per arm between Baseline and Week 48 visits.
Time Frame: Baseline and Week 48
Population: Values included for all enrolled participants excluding participants with confirmed virologic failure or those missing values due to early withdrawal, loss to follow-up or other error.
Measure: Mean (Standard Deviation); unit: percentage of prescribed doses
Arm/Group | Control Arm | Intervention Arm No.1 | Intervention Arm No.2 | Total
Number analyzed (Participants) | 12 | 13 | 10 | 35
percentage of prescribed doses
  3 Day Adherence Recall at Baseline | 100 (0) | 97.5 (9.2) | 96.7 (10.4) | 98.1 (7.8)
  3 Day Adherence Recall at Week 48 | 100 (0) | 97.5 (9.2) | 95.0 (15.8) | 97.6 (10)
  Change in 3 Day Adherence Recall | 0 (0) | 0 (13.5) | -1.7 (19.9) | -0.5 (13)

4. Secondary Outcome: Change in Quality of Life From Baseline to 48 Weeks of Study Treatment
Description: Quality of Life was measured by self report using a standardized scale, where 0 is death and 100 is perfect health. The baseline measure was obtained prior to initiation of study treatment arm. The week 48 measure captures Quality of Life by self report at 48 weeks of study treatment.
Time Frame: baseline and 48 weeks
Population: Data for all participants assigned to a study treatment was analyzed except data for participants that did not have both baseline and week 48 data, including early withdrawal, virologic failure, loss to follow-up or missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Arm | Intervention Arm No.1 | Intervention Arm No.2 | Total
Number analyzed (Participants) | 11 | 12 | 8 | 31
units on a scale
  Mean Quality of Life Score at Baseline | 92.9 (8.6) | 77.4 (16.1) | 82.5 (11.6) | 84.2 (14.1)
  Mean Quality of Life Score at Week 48 | 90.5 (11.1) | 78.2 (22.6) | 81.3 (17.5) | 83.3 (18.2)
  Change in Quality of Life | -2.5 (8.2) | 0.8 (20.0) | -1.3 (12.7) | -0.9 (14.4)

ADVERSE EVENTS:
Time Frame: 48 Weeks
Arm/Group | Control Arm | Intervention Arm No.1 | Intervention Arm No.2 | Total
Serious Adverse Events (participants affected / at risk) | 1/14 | 2/15 | 2/14 | 5/43
Other Adverse Events (participants affected / at risk) | 9/14 | 13/15 | 13/14 | 35/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=14) | Intervention Arm No.1 (N=15) | Intervention Arm No.2 (N=14) | Total (N=43)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hospitalization due to asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hospitalization for Recurrent Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=14) | Intervention Arm No.1 (N=15) | Intervention Arm No.2 (N=14) | Total (N=43)
hypertophy of tonsils (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ECG changes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
palpitations without chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
eustacian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
visual disturbance (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
apthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
changes to bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
dental pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3) | 6 (6)
dry throat (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
feeling full upon awakening (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
GI disturbance (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
heart burn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
tooth abscess (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Nightsweats (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
weight gain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
influenza like illness (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
latent mycobacterium tuberculosis Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
scabies (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
STI (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
bone fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
facial laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
leg pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
lower extremity ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
lower extremity pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
popliteal cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2) | 6 (6)
insomnia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
light headedness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
paresthesias (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
vivid dreams (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Renal Calculus (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (2) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus Pressure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 3 (3) | 4 (5)
Abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 1 (1) | 3 (4)
Angular Chelitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cutaneous Sarcoidosis, worsening (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Groin Itch (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
loose nails - bilateral halux (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Skin Rash, unspecified (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Tinea Cruris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Substance Misuse (Social circumstances) | 1 (1) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes